CLINICAL TRIAL: NCT02077842
Title: Prophylactic Nasal Continuous Positive Airway Pressure in the Post-Anaesthesia Care Unit Following Elective Laparotomy for Bowel Surgery
Brief Title: Prophylactic nCPAP in the PACU Following Elective Laparotomy for Bowel Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, William McKay, Anesthesiologist, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-192
Record Dates: First submitted 2014-03-02; First posted 2014-03-04 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Pulmonary Atelectasis; Surgery
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal CPAP (Experimental): The experimental group will receive nasal continuous positive airway pressure at 10cmH20 for one hour in the Post Anesthetic Care Unit.
  Interventions: Device: Nasal Continuous Positive Airway Pressure
- Low Flow Oxygen (Active Comparator): The control group will receive standard therapy of low flow oxygen via simple mask at 8 litres per minute.
  Interventions: Device: Low Flow Oxygen

INTERVENTIONS:
Device: Nasal Continuous Positive Airway Pressure — Nasal continuous positive airway pressure at 10 cmH2O
  Other Names: Resmed, VPAP III ST-A, manufactured by ResMed LTD
  Arms: Nasal CPAP
Device: Low Flow Oxygen — Low flow oxygen delivered via face mask at 8 litres per minute
  Arms: Low Flow Oxygen

SUMMARY:
The purpose of this study is to determine whether prophylactic nasal continuous positive airway pressure (nCPAP) in the post-anaesthesia care unit (PACU) improves post-operative pulmonary function following elective bowel surgery. The investigators hypothesize that one hour of nCPAP in the PACU will result in a higher partial pressure of arterial oxygen (PaO2) when compared to the standard treatment of low flow oxygen applied by face mask.

DETAILED DESCRIPTION:
Post-operative pulmonary complications, such as hypoxemia, pneumonia and respiratory failure, occur in 5-10% of patients following abdominal surgery. These post-operative pulmonary complications result in increased morbidity, mortality, ICU admission, length of hospital stay and resource use.

CPAP has shown to be an effective treatment for hypoxemia following abdominal surgery. It decreases atelectasis formation the risk of pneumonia. Application of nCPAP to treat hypoxemic respiratory failure following thoraco-abdominal surgery has shown to decrease endotracheal intubation.

Nasal CPAP has shown to be effective prophylaxis following elective cardiac and thoraco-abdominal aortic surgery. It reduces the incidence of hypoxemia, pneumonia, re-intubation and re-admission to the ICU. It has also shown to decrease the length of hospital stay.

The use of nCPAP immediately post-operatively in the PACU following abdominal surgery has not been evaluated. Nasal CPAP is better tolerated than full face mask CPAP. It allows for effective clearance of respiratory secretions, improved communication and decreases claustrophobic sensation. The PACU is a transition period from general anaesthesia into the post-operative recovery phase. During this time, residual anaesthetic causes decreased level of consciousness and sub-optimal respiratory effort. Reversal agent for neuromuscular blockade has often not reached its peak effect. Inadequate pain control may further decrease respiratory effort. This transition period may be when maximal atelectasis of alveolar lung units occurs. This time period may be optimal for the application of nCPAP for prophylaxis against hypoxemia. It may improve post-operative pulmonary function which could decrease post-operative morbidity, mortality, length of hospital stay and resource use.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo laparotomy for elective bowel surgery

Exclusion Criteria:

* age < 18 years
* postoperative admission to the intensive care unit
* a history of allergy/intolerance to Ametop

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Alveolar-arterial oxygen gradient | 1 hour after admission to the Post Anesthetic Care Unit
  The difference in the alveolar-arterial oxygen gradient between group administered nasal continuous positive airway pressure at 10cmH20 for one hour and group administered low flow oxygen by face mask at 8 litres per minute for one hour following elective bowel surgery

SECONDARY OUTCOMES:
Number of Participants Requiring Reintubation | 2 weeks
Number of Participants Requiring Admission to the Intensive Case Unit | 2 weeks
Length of Stay in Hospital | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William McKay, M.D., Principal Investigator — Faculty
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Zarbock A, Mueller E, Netzer S, Gabriel A, Feindt P, Kindgen-Milles D. Prophylactic nasal continuous positive airway pressure following cardiac surgery protects from postoperative pulmonary complications: a prospective, randomized, controlled trial in 500 patients. Chest. 2009 May;135(5):1252-1259. doi: 10.1378/chest.08-1602. Epub 2008 Nov 18. PMID 19017864
- [Background] Kindgen-Milles D, Muller E, Buhl R, Bohner H, Ritter D, Sandmann W, Tarnow J. Nasal-continuous positive airway pressure reduces pulmonary morbidity and length of hospital stay following thoracoabdominal aortic surgery. Chest. 2005 Aug;128(2):821-8. doi: 10.1378/chest.128.2.821. PMID 16100174
- [Background] Ferreyra GP, Baussano I, Squadrone V, Richiardi L, Marchiaro G, Del Sorbo L, Mascia L, Merletti F, Ranieri VM. Continuous positive airway pressure for treatment of respiratory complications after abdominal surgery: a systematic review and meta-analysis. Ann Surg. 2008 Apr;247(4):617-26. doi: 10.1097/SLA.0b013e3181675829. PMID 18362624